CLINICAL TRIAL: NCT04797117
Title: Analytical Validation of the abioSCOPE Device With a PSP Test: Point-of-Care Precision, Sample Type Comparison and Sample Stability
Acronym: AB-PSP-005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Abionic SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI21_0003 (AB-PSP-005)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Sepsis
Keywords: In Vitro Diagnostic Device; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sample (Other): The blood samples for the study for each patient will be collected in the form of additional tubes.
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — The blood samples for the study for each patient will be collected in the form of additional tubes.
  * either 1 tube of blood of 4 ml and 2 tubes of blood of 10 ml once a day for 1 or 2 days maximum (or 48 ml maximum) during his hospitalization
  * either 2 tubes of 10 ml or 20 ml maximum once during his hospitalization.

SUMMARY:
Abionic SA has developed a novel point-of-care (POC) platform, the abioSCOPE, and an in vitro diagnostic kit for the quantification of the pancreatic stone protein (PSP) to be analyzed specifically with the abioSCOPE® device. This test is intended to be used to aid in the early recognition of sepsis. The test is extremely easy to use and has a total turnaround time of approximately 8 minutes. This test uses only 30 microliters of K2/K3-EDTA anticoagulated whole blood or plasma. Results are quantitative (ng/ml). The product is for Investigational Use Only in the US and bears CE-marking. It is commercially available in selected European and non-European countries. The test has also been clinically validated in a multicentric, prospective, observational study performed (AB-PSP-001, clinicaltrials.gov identifier NCT03474809).

The main goals of this study are to evaluate certain analytical performances components of this product in a point-of-care environment, in particular the precision, sample type comparability and specimen stability of the product. Such data will support regulatory filing of a US FDA 510(k) premarket notification file and of a European IVD Regulation technical file to continue product commercialization in 2022, when this novel regulation will be effective.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated written informed consent by patient or close / family / trusted person prior to any mandatory study-specific procedures, sample collection, or analysis
* Male or female, 18 years of age or older;
* Hospitalized patient;
* Covered by a social security scheme.

Exclusion Criteria:

* Subject suffering from a hematological pathology (coagulation disorder, severe anemia) that could interfere with the blood draw procedure;
* Subject under juridical protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Precision variance components | Day 1
  coefficient of variation, expressed in percent, for the different variance components, are determined
Sample type comparison | Day 1
  pairwise comparability of test results when performed with K2-EDTA anticoagulated venous whole blood or K2-EDTA anticoagulated venous plasma, represented as percent recovery of whole blood compared to plasma, as well as scatter plots with Weighted Deming and Passing Bablok Regression, and bias plots.
Sample stability | Day 1
  Scatter plot and bias plot of PSP values versus storage time or freeze and thaw cycles, as well linear least square regression analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No